CLINICAL TRIAL: NCT04772144
Title: Smoking Cessation After a Cardiovascular Disease Event With Hospital-based Nurse-coordination and Further Follow-up Care in Lifestyle Centres With Free Cessation Aids - an Interdisciplinary Randomized Pilot Study
Brief Title: Nurse-led Smoking Cessation With Further Follow-up in Lifestyle Centres - a Randomized Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vestre Viken Hospital Trust (Other)
Collaborators: University of Oslo (Other); Norwegian Directorate of Health (Other Government); Oslo University Hospital (Other); Norwegian Institute of Public Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: REK 202686
Record Dates: First submitted 2021-01-07; First posted 2021-02-26 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Smoking Cessation; Smoking Behaviors; Nurse's Role; Cardiovascular Diseases
MeSH Terms: conditions — Smoking Cessation; Smoking; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: patients were randomized to an in-hospital nurse-led smoking cessation intervention with prescription of free cessation aids and systematic referrral to healthy life-centeres or usual care
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Behavioral: behavioural and cessation aids
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: behavioural and cessation aids — information, motivational interview, refferal to healty life-centers, free cessation aids
  Arms: Intervention group

SUMMARY:
The purpose of this randomized controlled pilot study is to test whether an in-hospital nurse-led smoking cessation intervention increases the refferal rate to healty life-centers in the municipalities. We will also describe the proportion who succeed in quitting smoking between the intervention group and the control group and obtain new knowledge about the patient and system factors of importance for participation to healty life-centers and for successful and unsuccessful smoking cessation.

ELIGIBILITY:
Inclusion Criteria (all):

* Age> 18 years and smokes at least 1 cigarette daily
* Hospitalized with a cardiovascular event (i.e. myocardial infarction, heart failure, unstable or stable angina, achyarrhythmias, bradyarrhythmias, carotid stenosis or claudication with need for peripheral revascularization)
* Sign informed consent and is expected to participate according to ICH / GCP

Exclusion Criteria (none of these):

* Does not meet the criteria to participate in the pilot project, i.e. patients who do not usually live or work in the Vestre Viken catchment area
* Chronic renal failure stage 4 or known allergic reaction to varenicline

  . Any condition (e.g. psychosis, alcohol abuse, dementia) or situation that may pose a significant risk to the participant, confuse the results or make participation unethical
* Lack of Norwegian and English knowledge
* Short life expectancy (<12 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Differences in participation rate at healthy life-centers between the intervention group and the control group measured by telephone interview with personnell at the healthy life-centers | 8-12 weeks after randomization
  Differences in participation rate at healthy life-centers between the intervention group and the control group measured by telephone interview with personnell at the healthy life-centers
Differences in use of smoking cessation aids between the intervention group and the control group | 8-12 weeks after randomization
  Differences in use of smoking cessation aids between the intervention group and the control group measued by patient self-report and collected from the prescription mediator in the hospital record

SECONDARY OUTCOMES:
Difference in point prevalence of smoke-free (no cigarettes last 7 days) after 6 months | 12 weeks after randomization
  Difference in point prevalence of smoke-free (no cigarettes last 7 days) after 6 months measured with self-reported questionnaires according to the Russell Standard
Difference between the groups in proportion who quit smoking between the groups | 12 weeks after randomization
  Difference between the groups in proportion who quit smoking between the groups measured by the level of carbon monoxide in the exhaled air

CONTACTS AND LOCATIONS:
Overall Officials: John munkhaugen, MD, PhD, Principal Investigator — Vestre Viken Trust, Drammen hospital
Locations (1):
- Drammen Hospital, Drammen, Akershus, Norway